CLINICAL TRIAL: NCT05857813
Title: Establishment of Social Skills Training Group in Adolescents With Autism Spectrum Disorder and Effectiveness Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202109033RIND
Record Dates: First submitted 2023-04-13; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASD teens and their caregiver (Experimental): Teens: (1) aged 11-20 years, currently enrolled in school between the sixth grade of elementary school and the third year of high school; (2) with a clinical diagnosis of ASD from a licensed mental health or medical professional based on DSM-5; (3) experiencing social difficulties as reported by parents in a structured intake interview; (4) scored ≧ 26 on the caregiver-reported Autism Spectrum Quotient (AQ), indicating clinical impairment associated with ASD (5) demonstrating verbal fluency in Chinese (6) with a full-scale IQ > 70 on WAIS-IV; (7) with motivation to participate in the intervention; (8) with a caregiver who was fluent in Chinese and willing to participate as a social coach in the study.
  Parents: (1) demonstrating verbal fluency in Chinese (2) with motivation to participate in the intervention and assist their children to do the homework assignments.
  Interventions: Behavioral: Program for the Education and Enrichment of Relational Skills (PEERS®)

INTERVENTIONS:
Behavioral: Program for the Education and Enrichment of Relational Skills (PEERS®) — developed at the University of California, Los Angeles (E. A. Laugeson & F. Frankel, 2010). This is a parent-assisted, manualized social skills training program that addresses crucial areas of social functioning for adolescents. Psycho-education and cognitive-behavioral therapy techniques are employed to help adolescents develop ecologically valid skills for making and maintaining friendships.

SUMMARY:
Autism spectrum disorders (ASD) is a neurodevelopmental disorder characterized by persistent deficits in social communication and social interaction across multiple contexts, and the presence of restricted, repetitive behavior and interests, affecting 1 in 68 children. Although atypical social deficits onset in early childhood, their social relationships with peers may remain a challenge or even worsen for individuals with ASD throughout the school years and beyond, as social contexts increase in complexity and pose higher social expectations.

ELIGIBILITY:
Inclusion Criteria:

* aged 11-20 years, currently enrolled in school between the sixth grade of elementary school and the third year of high school
* with a clinical diagnosis of ASD from a licensed mental health or medical professional based on DSM-5
* experiencing social difficulties as reported by parents in a structured intake interview
* scored ≧ 26 on the caregiver-reported Autism Spectrum Quotient (AQ), indicating clinical impairment associated with ASD
* demonstrating verbal fluency in Chinese
* with a full-scale IQ > 70 on WAIS-IV
* with motivation to participate in the intervention;
* with a caregiver who was fluent in Chinese and willing to participate as a social coach in the study.

Exclusion Criteria:

* a history of major mental illness (e.g., bipolar affective disorder, schizophrenia, or psychosis) or neurological diseases that might hinder participation in the treatment
* visual impairment and/or hearing impairment that would preclude participation in group-based social activities.

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-07-12 (Estimated); Study Completion 2027-07-12 (Estimated)

PRIMARY OUTCOMES:
Autism Diagnostic Interview-Revised (ADI-R) | 7 weeks
  Interview with caregiver of autistic participants. Total of 93 items coding from 1 to 9. Higher the score, worse the syptom
The Autism Diagnostic Observation Schedule (ADOS) | 7 weeks
  Observe the autistic participant during the interview. the examinee's condition is classified as autism spectrum if the combined score across two domains of social interaction and communication is ≥7, and as autism if the combined score is ≥12. In Module 2, a combined score of ≥8 corresponds to autism spectrum, and a combined score of ≥12 corresponds to autism
Autism Spectrum Quotient (AQ) | 7 weeks
  50 statement scoring from 1 to 4. higher the score, worse the syptom
Friendship Quality Scale (FQS) | 7 weeks
  23 questions scoring from 1 to 5. Higher the score, better the quality of friendship
The Assessing Emotions Scale (AES) | 7 weeks
  score range from 33 to 165. higher the score, better the emotional intelligence
Social Responsiveness Scale (SRS) | 7 weeks
  65 questions range from 1 to 4. higher the score, worse the symptom.
Social Adjustment Inventory for Children and Adolescents (SAICA) | 7 weeks
  17 scenarios scoring from 1 to 4. Higher the score, better the capability
Quality of Play Questionnaire (QPQ) | 7 weeks
  10 questions scoring from 0 to 3. Higher the score, worse the quality of play. Also, asked for frequency and number of participant in the play
Test of Adolescents Social Skills Knowledge (TASSK) | 7 weeks
  score range from 0 to 22. Higher the score, greater the knowledge of taught social skills
Empathy Quotient (EQ) | 7 weeks
  60 questions score from 0 to 3. Higher the score, greater the empathy
Friendship Questionnaire (FQ) | 7 weeks
  score from 0 to 135. higher the score, the more enjoyment of friendship

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan